CLINICAL TRIAL: NCT06042465
Title: Investigation on the Efficacy Between TCM Treatment Using Acupuncture and Tui-na Manipulation With Physiotherapy on Patellofemoral Pain Syndrome
Brief Title: Investigation on Efficacy Between TCM Treatment Using Acupuncture and Tui-na With Physiotherapy on Patellofemoral Pain Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hong Kong Baptist University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ACAO/L53/AY/2018
Record Dates: First submitted 2023-08-07; First posted 2023-09-18 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-03

CONDITIONS: Patellofemoral Pain Syndrome; Acupuncture; Physiotherapy
MeSH Terms: conditions — Patellofemoral Pain Syndrome | interventions — Acupuncture Therapy; Physical Therapy Modalities

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TCM group (Experimental): As decided and performed by the registered Chinese Medicine Practitioners (CMP) on standardized treatment method
  Interventions: Other: acupuncture and Tui-na manipulations
- PT group (Experimental): As decided and performed by physiotherapist of HKBH on standardized treatment method
  Interventions: Other: Physiotherapy
- Educational Group (No Intervention): Included patients in this group are provided with educational talk on knee health protection. Patients are advised with daily-life protection on their PFPS. Questionnaire assessments are performed to assess the healthy situation of their PFPS.

INTERVENTIONS:
Other: acupuncture and Tui-na manipulations — i. Patients in supine position with knee elevated 20-30 degrees bending using a pillow below.
  ii. Acupuncture needle using 0.25 mm diameter and 1.5-inch length. iii. Choose 'A shi point' to inject the acupuncture needles. iv. Inject 4 acupuncture needles respectively at the upper, lower, lateral and medial edge of the patella, along the medial and lateral edge at the posterior surface of patella.
  v. Connect the needles with electro-therapy, selecting high frequency and strength that the patients have sensation and acceptable. Time duration is 30 minutes each time. Infra-radiation is provided and warm above the treatment region.
  vi. Tui-na manipulations using the method of 'Tui-na'. Time duration is 2-5 minutes. Patella is pushed up and elevated during treatment.
  vii. No external herbal medicine for TCM group , other medication such as painkiller is required to record
  Arms: TCM group
Other: Physiotherapy — i. Total 12 sessions of physiotherapy for 8 weeks training; ii. Treatment: Closed kinetic chain exercises program will be used when appropriate, which include:
  1. Mini walk squat exercise
  2. Forward step up
  3. Lateral step up
  4. Terminal knee extension
  5. Knee taping
  6. Unstable base training
  7. Pain control
  8. Manual Therapy Each session will approximately cost each patient 1 hours' time. There is no Chinese medicine is allowed for PT group , other medication such as painkiller is required to record.
  Arms: PT group

SUMMARY:
Knee pain is one of common pain-causing diseases and it affects patients' mobility which in turn seriously affects the quality of patients' life. The most common cause of knee pain results from the inflammation occurred at the patello-femoral joint of the anterior knee. It is now commonly recognized as Patello-femoral pain syndrome (PFPS). It is categorized as anterior knee pain.

The exact pathogenesis of PFPS is still not clear but both Traditional Chinese Medicine (TCM) and Western Medicine (WM) have many treatment methods. Hence, it is important and meaningful to investigate the diagnosis and treatment in detail. Through reviewing the literature about PFPS, the investigators would like to achieve the following objectives in the study design. Under the principle of evidence-based medicine, the investigators compare the clinical effectiveness of TCM acupuncture and Tui-na manipulations treatment with the physiotherapy on the PFPS management. The study is to determine whether which are effective in improving knee function and lessening the pain in PFPS patients.

DETAILED DESCRIPTION:
The target sample size will be 180 patients approximately, each group namely Traditional Chinese Medicine (TCM)/ Physiotherapy (PT)/ Education group respectively will contain minimum 60 patients respectively. Patients are initially screened with questionnaire implying the PFPS scouring system. Patients will be recruited and firstly screened from Chinese Medicine Practitioner (CMP). Then the secondary screening will be conducted by the WM practitioner in Hong Kong Baptist Hospital (HKBH) to confirm diagnosis and enrollment based on the inclusion and exclusion criteria. X-ray imaging diagnosis and reporting are done in HKBH.

The investigators will design a randomized controlled trial, compared with TCM group and PT group. Patients are requested to sign a consent form before entering the washout period for 2 weeks before they start their interventions. TCM group will receive acupuncture and Tui-na. PT group will receive physiotherapy training. Patients will be treated twice a week and rest on 3rd and 6th week. Total 12 sessions treatments within 8 weeks. The investigators set up a control group named "education group", the control group will be used to compare with the other two groups. Included patients in this group are provided with educational talk on knee health protection. Patients are advised with daily-life protection on their PFPS. After 8 weeks of control intervention, patients are given with treatment same as TCM group or PT group in 1:1 basis. Phone-follow up will start from 3-month after the treatment.

Statistical analysis will be performed using the Social Science Statistics Package (SPSS) for Windows version. The investigators are going to (1) analysis of the PFPS diagnostic criteria; (2)Comparison between the questionnaire and examinations before and after the treatment intervention.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70, male and female, knee pain as main complaint;
2. Diagnosed as PFPS using our diagnostic standard;
3. Knee pain for more than 1 month;
4. Patients could be able to finish all questionnaires, treatment;
5. Insidious onset of symptoms unrelated to a traumatic incident and persistent for at least 6 weeks;
6. Able to cooperate with questionnaires, examination and treatment and follow-up cycles;
7. Agree to receive regular Chinese medicine diagnosis and assist in the designated examinations in the study.
8. Agree to record physical condition indicators and report the situation at each follow-up consultation.
9. During the entire plan period, the subjects must agree not to use any type of Chinese medicine health care products until the end of the trial.

Exclusion Criteria:

1. Age below 18 and above 70; Patients with Body Mass Index (BMI)≧30;
2. Patients with acute traumatic bone fracture, dislocation or acute soft tissue injury at knee joint;
3. Patients with infections at knee joint;
4. Patients with non-specific inflammation at knee joint and rheumatoid disease;
5. Patients with ostomy or other tumor related;
6. Patients with knee pain but not anterior knee pain, e.g. meniscal or other intra articular pathologic condition, cruciate or collateral ligament cases, patella subluxation or dislocation, previous surgery in the knee and hip joints, knee and hip joint osteoarthritis, any conditions affect muscle strength like diabetes mellitus or rheumatoid arthritis；
7. Patients with patellar tendon inflammation or Osgood-Schlatter Disease;
8. Any psychiatric disorder;
9. Pregnancy;
10. Patients with severe disease such as immune disease, genetic disease and severe coronary vascular disease;
11. Patients receive any other treatment such as physiotherapy or acupuncture after washout period.
12. If participants are incompetent in giving consent .

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-10-18 (Actual); Primary Completion 2023-10-18 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Effectiveness Measurement | 3 months
  The expected outcomes are both interventions have effectiveness on curing the PFPS. Traditional Chinese Medicine group and Physiotherapy group have better effectiveness than control group in treating PFPS. By according to the Visual Analogue Scale score and the before and after evaluation form, it indicates whether the pain condition has improved.
  (Visual Analogue Scale will be indicated from 0 to 10. Which 0 stand for no pain at all and 10 marks stand for the worst pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Kevin Yue Kin Man, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No